CLINICAL TRIAL: NCT04553406
Title: A Randomized, Partially Blinded, Placebo- and Comparator-Controlled, Multicenter, Phase 2a, Dose Ranging, Proof-of-Concept Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SPR720 as Compared With Placebo or Standard of Care for the Treatment of Patients With Mycobacterium Avium Complex (MAC) Pulmonary Disease
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of SPR720 for the Treatment of Patients With Mycobacterium Avium Complex (MAC) Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision pending resolution of clinical hold with FDA
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR720-201
Record Dates: First submitted 2020-09-01; First posted 2020-09-17 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-11

CONDITIONS: Mycobacterium Avium Complex; Non-tuberculous Mycobacterium Pulmonary Disease
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment Arms 1 to 3 are masked while Treatment Arm 4 is open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SPR720 low dose (Experimental): SPR720 500 mg administered orally once daily for 28 days.
  Interventions: Drug: SPR720
- SPR720 high dose (Experimental): SPR720 1000 mg administered orally once daily for 28 days.
  Interventions: Drug: SPR720
- Placebo (Placebo Comparator): Placebo administered orally once daily for 28 days
  Interventions: Drug: Placebo
- Standard of Care (SOC) (Active Comparator): Standard of Care regimen per the Investigator's discretion.
  Interventions: Drug: Open-label Standard of Care

INTERVENTIONS:
Drug: SPR720 — Capsules for oral administration
  Arms: SPR720 high dose; SPR720 low dose
Drug: Placebo — Capsules for oral administration
  Arms: Placebo
Drug: Open-label Standard of Care — Standard of Care regimen is at the Investigator's discretion; recommended 2-drug or 3-drug SOC, consisting of either:
  * Clarithromycin 500-1000 mg, plus ethambutol hydrochloride (HCl) 15 mg/kg orally once daily or
  * Azithromycin 250-500 mg plus ethambutol HCl 15 mg/kg orally once daily.
  Optional rifampin 600 mg or rifabutin 300 mg orally once daily may be added to the SOC regimen for up to 28 days.
  Arms: Standard of Care (SOC)

SUMMARY:
To evaluate the pharmacokinetics (PK) of SPR719, the active moiety, generated from the orally (po) administered SPR720 prodrug in a patient population with nontuberculous mycobacteria pulmonary disease (NTM-PD)

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of NTM-PD due to MAC
* Had at least 1 prior positive culture (sputum or bronchoalveolar lavage) positive for MAC in the previous 6 months
* Has an induced sputum culture at screening positive for MAC by at least one of the following methods performed by the microbiology laboratory: quantitative culture on solid agar or growth on liquid media (MGIT)
* Is either treatment naïve and has not received any prior treatment for MAC, OR if previously treated for MAC, has culture evidence of persistent, recurrent, or relapsed disease and has been off therapy for at least 6 months
* In the opinion of the Investigator, is ready to initiate treatment (treatment naïve) or reinitiate treatment (previously treated) within the next 3 months, and for whom a delay, in order to participate in a placebo-controlled clinical trial, is considered reasonable and clinically acceptable
* Had clinical signs and symptoms within the 6 weeks before the date of consent that are consistent with NTM-PD with at least two of the following:

  1. chronic cough
  2. fatigue
  3. frequent throat clearing
  4. shortness of breath (dyspnea)
  5. coughing up of blood (hemoptysis)
  6. excessive mucus (sputum) production
  7. fever
  8. night sweats
  9. loss of appetite
  10. unintended weight loss
  11. wheezing
  12. chest pain
* Has a measured forced expiratory volume in 1 second (% predicted FEV1) ≥30% on pulmonary function test within 3 months prior to consent
* Has a chest radiograph (CXR) or computed tomography (CT) scan within 6 months prior to consent with findings consistent with NTM-PD. If no CXR or CT scan is available, a CXR or CT scan should be performed at screening to confirm eligibility.
* Other inclusion criteria per protocol

Exclusion Criteria:

* Has disseminated or extrapulmonary NTM
* Has end-stage NTM-PD or treatment-refractory NTM-PD and is unlikely to respond to protocol-specified SOC treatment
* Had isolation on sputum cultures of any species of Mycobacterium other than a species included in MAC within the past 6 months
* Had prior isolation of MAC with macrolide resistance
* Has received any systemic (oral or IV) or inhaled antibiotic with activity against MAC between consent and randomization
* Has a potentially confounding underlying pulmonary disease, including but not limited to cystic fibrosis, active pulmonary malignancy (primary or metastatic), NTM-hypersensitivity disease pneumoconiosis, or another advanced lung disease with a % predicted FEV1<30%
* Other exclusion criteria per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — Spero Therapeutics Inc
Locations (9):
- United States (9):
  - Medical Facility, Altamonte Springs, Florida
  - Medical Facility, Atlantis, Florida
  - Medical Facility, Clearwater, Florida
  - Medical Facility, Kissimmee, Florida
  - Medical Facility, West Palm Beach, Florida
  - Medical Facility, Charlotte, North Carolina
  - Medical Facility, Mooresville, North Carolina
  - Medical Facility, Winston-Salem, North Carolina
  - Medical Facility, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 participants were planned to be enrolled across 4 treatment groups. As a result of early discontinuation of the study, only 2 treatment groups were initiated, with 1 participant enrolled in each group.
Groups:
- SPR720 500 mg: SPR720 500 mg administered orally once daily for 28 days.
Period: Overall Study
Arm/Group | SPR720 500 mg | Placebo
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Study Discontinuation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPR720 500 mg | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of SPR719
Description: SPR719 is the active moiety of the prodrug SPR720. Blood samples were planned to be taken at a subset of study sites in order to conduct intensive pharmacokinetic (PK) evaluation.
Time Frame: Day 1 and Day 28 pre-dose and 1, 2, 4, 8, 12, and 24 hours post-dose
Population: No participants were enrolled at study sites that were conducting intensive PK evaluations.
Arm/Group | SPR720 500 mg
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of SPR719
Time Frame: Day 1 and Day 28 pre-dose and 1, 2, 4, 8, 12, and 24 hours post-dose
Population: No participants were enrolled at study sites that were conducting intensive PK evaluations.
Arm/Group | SPR720 500 mg
Number analyzed (Participants) | 0

3. Primary Outcome: Area Under the Concentration-time Curve From Zero to Tau, Where Tau is the Dosing Interval (AUC0-tau) for SPR719
Time Frame: Day 1 and Day 28 pre-dose and 1, 2, 4, 8, 12, and 24 hours post-dose
Population: No participants were enrolled at study sites that were conducting intensive PK evaluations.
Arm/Group | SPR720 500 mg
Number analyzed (Participants) | 0

4. Primary Outcome: Accumulation Ratio of SPR719
Time Frame: Day 1 and Day 28 pre-dose and 1, 2, 4, 8, 12, and 24 hours post-dose
Population: No participants were enrolled at study sites that were conducting intensive PK evaluations.
Arm/Group | SPR720 500 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product, which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational/experimental) product, whether related to this product or not. This includes any newly occurring event or previous condition that has increased in severity or frequency since starting active or randomized treatment.
  The Investigator assessed the intensity for each AE reported during the study using the latest version of the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, as Mild, Moderate, Severe, Life-threatening, or Death.
Time Frame: From first dose of study drug (Day 1) up to 28 days after last dose (56 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 1 | 1
Participants
  All TEAEs | 1 | 1
  Mild TEAEs | 1 | 1
  Moderate TEAEs | 0 | 0
  Severe TEAEs | 0 | 0
  TEAEs leading to discontinuation of study drug | 0 | 0
  TEAEs leading to discontinuation from study | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Meaningful Change in Physical Examination Findings
Description: Full physical examination were conducted on Day 1 and 28 days after last dose (Day 56) and included, at a minimum, assessment of the following systems: skin, head, ears, eyes, nose and throat, respiratory system, cardiovascular system, gastrointestinal system, neurological condition, blood and lymphatic systems, and the musculoskeletal system. Symptom-directed physical examinations were conducted at study visits on Days 7, 14, 21, and 28.
Time Frame: Days 1, 7, 14, 21, 28, and 56
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Who Received Any Concomitant Medication During the Study
Time Frame: Day 1 to Day 56
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

8. Secondary Outcome: Changes From Baseline in Laboratory Tests
Time Frame: Days 1, 7, 14, 21, 28, and 56
Population: Individual laboratory test results are not reported in order to protect patient confidentiality.
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Out-of-normal Range Laboratory Tests
Description: Clinical laboratory tests included serum chemistry, hematology, coagulation tests, and urinalysis. The investigator determined whether any changes in laboratory values were clinically significant based on the condition of the participant and the extent and duration of the deviation from the reference range.
Time Frame: Days 1, 7, 14, 21, 28, and 56
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 1 | 1
Participants
  Clinical chemistry | 0 | 0
  Hematology | 0 | 0
  Coagulation tests | 0 | 0
  Urinalysis | 0 | 0

10. Secondary Outcome: Shifts From Baseline in Selected Laboratory Tests Using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Shift Categories
Time Frame: Days 1, 7, 14, 21, 28, and 56
Population: No participants had out-of-range laboratory test results hence shift tables could not be created.
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Changes From Baseline in Vital Sign Measurements
Description: Vital signs measurements included systolic and diastolic blood pressure, pulse, temperature, and respiratory rate.
Time Frame: Days 1, 7, 14, 21, 28, and 56
Population: Individual vital sign measurement results are not reported in order to protect patient confidentiality.
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram Findings
Description: Standard 12-lead electrocardiogram (ECG) assessments included heart rate, cardiac rhythm, PR interval, RR interval, QRS interval, QT interval and QTC interval. Clinical significance was determined by the investigator.
Time Frame: Days 1, 14, 28, and 56
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | SPR720 500 mg | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study up to 28 days after last dose (56 days).
Arm/Group | SPR720 500 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPR720 500 mg (N=1) | Placebo (N=1)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish the results prior to the first multi-site publication. If there is no multi-site publication within 18 months after Trial completion the PI may publish results from the trial, subject to the following. PI will submit proposed Publication to Sponsor 60 days prior to submission of the Publication. PI will, at Sponsor's request, delay such Publication for up to 90 days for Sponsor to obtain appropriate intellectual property protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04553406/Prot_SAP_000.pdf